CLINICAL TRIAL: NCT07337941
Title: The Effects of Menstrual Cycle Phase and Virtual Reality on Preoperative Anxiety
Brief Title: Menstrual Cycle Phase and Virtual Reality on Preoperative Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Gamze Küçükosman, Principal Investigator, Department of Anesthesiology and Reanimation, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021/21 VR
Record Dates: First submitted 2025-12-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: American Society of Anesthesiologists (ASA) I-II Risk Groups; the Follicular (Days 1-12 From Last Menstruation) or Luteal (Days 20-24) Phase of the Menstrual Cycle; Aged 18-55
Keywords: Virtual Reality; Preoperative Anxiety; Menstrual Cycle Phase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Gorup 2: Luteal Phase + No VR (Placebo Comparator): The 15-minute immersive virtual reality video, which offered both visual and auditory stimuli, was not shown.
  In the preoperative period, heart rate and mean arterial pressure values were recorded at baseline, and at 5, 10, and 15 minutes over a 15-minute period. Participants were asked to complete the STAI I-II anxiety scales only once.
  Interventions: Other: State-Trait Anxiety Inventory (STAI I-II); Other: The decision for a 15-minute preoperative observation without visual and auditory experience depends on the phase of the menstrual cycle and group assignment.
- Group 3: Follicular Phase + Virtual Reality (VR) (Active Comparator): 15-minute immersive virtual reality video providing both visual and auditory stimuli .Baseline and 5th, 10th, and 15th minute heart rate and mean arterial pressure values were recorded during the viewing of the video. After the video, the headset was removed, and the patients were asked to complete STAI I-II again.
  Interventions: Other: 15-minute video providing a visual and auditory experience (Training Video); Other: State-Trait Anxiety Inventory (STAI I-II)
- Group 4: Follicular Phase + No VR (Placebo Comparator): The 15-minute immersive virtual reality video, which offered both visual and auditory stimuli, was not shown.
  In the preoperative period, heart rate and mean arterial pressure values were recorded at baseline, and at 5, 10, and 15 minutes over a 15-minute period. Participants were asked to complete the STAI I-II anxiety scales only once.
  Interventions: Other: State-Trait Anxiety Inventory (STAI I-II); Other: The decision for a 15-minute preoperative observation without visual and auditory experience depends on the phase of the menstrual cycle and group assignment.
- Group 1:Luteal Phase+ Virtual Reality (VR) (Active Comparator): 15-minute immersive virtual reality video providing both visual and auditory stimuli .Baseline and 5th, 10th, and 15th minute heart rate and mean arterial pressure values were recorded during the viewing of the video. After the video, the headset was removed, and the patients were asked to complete STAI I-II agai
  Interventions: Other: 15-minute video providing a visual and auditory experience (Training Video); Other: State-Trait Anxiety Inventory (STAI I-II)

INTERVENTIONS:
Other: 15-minute video providing a visual and auditory experience (Training Video) — Whether or not to watch a 15-minute video (Training Video) offering a visual and auditory experience, depending on the menstrual phase and group distribution.
  Arms: Group 1:Luteal Phase+ Virtual Reality (VR); Group 3: Follicular Phase + Virtual Reality (VR)
Other: State-Trait Anxiety Inventory (STAI I-II) — Anxiety levels are scored as "(1) not at all, (2) a little, (3) a lot, and (4) completely" on the STAI-I, while the STAI-II options are (1) almost never, (2) sometimes, (3) a lot, and (4) almost always. There are two types of statements on the scales: direct statements express negative emotions, while reverse statements express positive emotions. Two separate total score weights are calculated for each direct and reverse statement. The total score for reverse statements is subtracted from the total score obtained for direct statements. A predetermined and constant value is added to this number. 50 is added as a constant value to the number obtained for the STAI-I. For the STAI-II, this value is 35. The final value is the individual's anxiety score. Scores from both scales theoretically range from 20 to 80. A high score indicates a high level of anxiety.
Other: The decision for a 15-minute preoperative observation without visual and auditory experience depends on the phase of the menstrual cycle and group assignment. — The decision for a 15-minute preoperative observation without visual and auditory experience depends on the phase of the menstrual cycle and group assignment.
  Arms: Gorup 2: Luteal Phase + No VR; Group 4: Follicular Phase + No VR

SUMMARY:
This study aims to examine the effects of menstrual cycle phase and a virtual reality (VR) intervention on preoperative anxiety in female patients scheduled for septorhinoplasty surgery.

DETAILED DESCRIPTION:
This study was designed to evaluate the effects of menstrual cycle phases (follicular/luteal) and the use of virtual reality (VR) on preoperative anxiety levels and hemodynamic parameters in female patients scheduled for septorhinoplasty surgery. The study consisted of four groups: follicular phase with VR, follicular phase without VR, luteal phase with VR, and luteal phase without VR. All participants' preoperative anxiety levels were assessed using the State-Trait Anxiety Inventory (STAI I-II) and the Amsterdam Preoperative Anxiety and Information Scale (APAIS). In the VR groups, heart rate and mean arterial pressure were recorded at baseline and at 5, 10, and 15 minutes during the video session. This study aims to determine whether VR, as a non-pharmacological method, is an effective tool for managing preoperative anxiety.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I-II risk groups,
* scheduled for elective septorhinoplasty,
* either the follicular (days 1-12 from last menstruation) or luteal (days 20-24) phase of the menstrual cycle

Exclusion Criteria:

* if they did not speak Turkish
* in days 13-19 of their menstrual cycle,
* menstrual irregularities,
* undergone hysterectomy or bilateral salpingo-oophorectomy,
* drug allergies,
* psychiatric or cognitive dysfunction,
* epilepsy,
* claustrophobia,
* alcohol-substance dependence,
* blindness or deafness,
* revision septorhinoplasty.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 170 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Amsterdam Preoperative Anxiety and Information Scale (APAIS) Score | Preoperative (before VR or baseline)
State-Trait Anxiety Inventory (STAI-I/II) Score | Preoperative and Post-Intervention (after 15-minute video or control period)

SECONDARY OUTCOMES:
Heart Rate | At baseline, and at 5, 10, and 15 minutes during video viewing

CONTACTS AND LOCATIONS:
Locations (1):
- Gamze Küçükosman, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided